CLINICAL TRIAL: NCT03985878
Title: An Open-Label Safety, Tolerability, and Efficacy Study of Eteplirsen in Patients With Duchenne Muscular Dystrophy Who Have Completed Study 4658-102
Brief Title: A Study to Evaluate Safety, Tolerability, and Efficacy of Eteplirsen in Participants With Duchenne Muscular Dystrophy (DMD) Who Have Completed Study 4658-102 (NCT03218995)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Participants were either transitioned to a post-trial access program or another Sarepta study, or they declined further treatment. There are no safety concerns with Eteplirsen.
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4658-102-OLE; 2019-000337-39 (EudraCT Number)
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Results first posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-07

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD; Duchenne; Eteplirsen; Dystrophy; Dystrophin; Exon Skipping; Exon 51; Ambulatory; Pediatric
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — eteplirsen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eteplirsen (Experimental): Participants will receive eteplirsen via IV infusions, once weekly, for up to 284 weeks.
  Interventions: Drug: Eteplirsen

INTERVENTIONS:
Drug: Eteplirsen — Eteplirsen IV infusion once weekly.
  Other Names: AVI-4658; EXONDYS 51; EXONDYS

SUMMARY:
The purpose of this extension study is to evaluate the ongoing safety and tolerability of additional treatment with eteplirsen administered once weekly by intravenous (IV) infusion in male participants with DMD who have successfully completed the 96-week eteplirsen Study 4658-102.

ELIGIBILITY:
Inclusion Criteria:

* Participant successfully completes 96 weeks of treatment in Study 4658-102.

Exclusion Criteria:

* Participant has a prior or ongoing medical condition that, in the Investigator's opinion, could adversely affect the safety of the participant, or make it unlikely that the course of treatment or follow-up would be completed, or impair the assessment of study results.

Other inclusion/exclusion criteria apply.

Ages: 2 Years to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (4):
- UZ-Gent, Ghent, Belgium
- Hopital Trousseau, Bâtiment lemariey, Paris, France
- Fondazione Policlinico Universitario Agostino Gemelli, UOC Neuropsichiatria Infantile, Rome, Italy
- UCL Great Ormond Street Institute of Child Health, Dubowitz Neuromuscular Centre, London, England, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In an effort to reduce clinical trial burden on participants while ensuring continued treatment if desired, pending commercial availability of eteplirsen, participants were either transitioned to a post-trial access program or another Sarepta study, or they declined further treatment.
Groups:
- Eteplirsen: Participants received eteplirsen via intravenous (IV) infusions, once weekly, for up to 162 weeks.
Period: Overall Study
Arm/Group | Eteplirsen
Started | 15
Received At Least 1 Dose Of Study Drug (Safety Set) | 15
Completed | 0
Not Completed | 15
Not completed — Transitioned to Another Sarepta Study | 2
Not completed — Study Terminated by Sponsor | 12
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Safety Set: all participants who received eteplirsen.
Groups:
- Eteplirsen: Participants received eteplirsen via IV infusions, once weekly, for up to 162 weeks.
Arm/Group | Eteplirsen
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.7 (1.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' section.
Time Frame: Up to 162 weeks
Population: Safety Set: all participants who received eteplirsen.
Measure: Number; unit: Participants
Arm/Group | Eteplirsen
Number analyzed (Participants) | 15
Participants | 15

2. Primary Outcome: Number of Participants Experiencing Death Due to Adverse Events
Description: A summary of all deaths regardless of causality is located in the 'Reported Adverse Events' section.
Time Frame: Up to 162 weeks
Population: Safety Set: all participants who received eteplirsen.
Measure: Number; unit: Participants
Arm/Group | Eteplirsen
Number analyzed (Participants) | 15
Participants | 0

3. Primary Outcome: Number of Participants Experiencing Adverse Events of Special Interest (AESIs)
Description: AESIs were defined as any AE that was of scientific and medical concern specific to study treatment, for which ongoing and rapid communication by the Investigator to the sponsor was appropriate. AESIs included findings potentially indicative of hepatic and renal abnormalities, hypersensitivity, and thrombocytopenia. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' section.
Time Frame: Up to 162 weeks
Population: Safety Set: all participants who received eteplirsen.
Measure: Number; unit: Participants
Arm/Group | Eteplirsen
Number analyzed (Participants) | 15
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 162 weeks
Description: Safety Set: all participants who received eteplirsen. In an effort to reduce clinical trial burden on participants while ensuring continued treatment if desired, pending commercial availability of eteplirsen, participants were either transitioned to a post-trial access program or another Sarepta study, or they declined further treatment.
Arm/Group | Eteplirsen
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eteplirsen (N=15)
Influenza (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eteplirsen (N=15)
Nasopharyngitis (Infections and infestations) | 8
Corona virus infection (Infections and infestations) | 7
Rhinitis (Infections and infestations) | 6
Enterobiasis (Infections and infestations) | 3
Influenza (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Foot and mouth disease (Infections and infestations) | 1
Genital infection fungal (Infections and infestations) | 1
Helminthic infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Molluscum contagiosum (Infections and infestations) | 1
Onychomycosis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Dental caries (Gastrointestinal disorders) | 2
Abdominal pain lower (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 9
Influenza like illness (General disorders) | 3
Gait disturbance (General disorders) | 2
Catheter site pain (General disorders) | 1
Catheter site swelling (General disorders) | 1
Chest pain (General disorders) | 1
Device dislocation (General disorders) | 1
Hyperpyrexia (General disorders) | 1
Infusion site extravasation (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 5
Fall (Injury, poisoning and procedural complications) | 5
Head injury (Injury, poisoning and procedural complications) | 3
Excoriation (Injury, poisoning and procedural complications) | 2
Face injury (Injury, poisoning and procedural complications) | 2
Scratch (Injury, poisoning and procedural complications) | 2
Skin abrasion (Injury, poisoning and procedural complications) | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1
Eye contusion (Injury, poisoning and procedural complications) | 1
Human bite (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Ecchymosis (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Keloid scar (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Headache (Nervous system disorders) | 6
Cognitive disorder (Nervous system disorders) | 1
Motor dysfunction (Nervous system disorders) | 1
Psychomotor hyperactivity (Nervous system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Ear pain (Ear and labyrinth disorders) | 2
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 1
Chalazion (Eye disorders) | 2
Eye pain (Eye disorders) | 1
Eye pruritus (Eye disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Weight gain poor (Metabolism and nutrition disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Dilatation ventricular (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Initial insomnia (Psychiatric disorders) | 1
Irritability (Psychiatric disorders) | 1
Chromaturia (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Myoglobinuria (Renal and urinary disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Urine albumin/creatinine ratio abnormal (Investigations) | 1

LIMITATIONS AND CAVEATS:
In an effort to reduce clinical trial burden on participants while ensuring continued treatment if desired, pending commercial availability of eteplirsen, participants were either transitioned to a post-trial access program or another Sarepta study, or they declined further treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There are agreements between the Principal Investigators and the Sponsor (or its agents) that restrict the PIs rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT03985878/Prot_SAP_000.pdf